CLINICAL TRIAL: NCT00894465
Title: A Randomized, Double-Blind, Placebo-Controlled Study Examining the Efficacy of Oral Midazolam in Reducing Anxiety in Children Undergoing Voiding Cystourethrogram
Brief Title: Midazolam Effect in Children Undergoing Voiding Cystourethrogram (VCUG)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Most pts requested to be treated with versed. It was difficult to randomize pts.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Society of Pediatric Urology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: HRPO # 06-0665
Record Dates: First submitted 2009-05-04; First posted 2009-05-07 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Vesicoureteral Reflux
Keywords: Midazolam; VCUG; Anxiety
MeSH Terms: conditions — Vesico-Ureteral Reflux; Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Versed (Experimental): Both patients who are VCUG naive and patients who have had a previous VCUG are given oral midazolam prior to undergoing the VCUG.
  Interventions: Drug: midazolam
- Placebo (Placebo Comparator): Both patients who are VCUG naive and patients who have had a previous VCUG are given an oral placebo prior to undergoing the VCUG.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: midazolam — Children are randomized to receive oral midazolam .5 mg/kg prior to undergoing VCUG
  Arms: Versed
Drug: placebo — Children are randomized to receive a placebo prior to undergoing VCUG
  Arms: Placebo

SUMMARY:
The purpose of this research is to validate the common administration of oral midazolam to children prior to voiding cystourethrogram (VCUG) to see if this will significantly decrease children's anxiety and make the experience less traumatic.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-6 years
* Toilet trained
* English speaking
* Already scheduled for VCUG

Exclusion Criteria:

* Allergic to midazolam
* Active UTI
* Known urethral stricture
* Known urethral reconstruction
* Has history of abnormal sensation in pelvic area
* Has history of sexual abuse
* Has severe developmental delay
* Has diagnosis of anxiety disorders

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Austin, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Versed | Placebo
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who signed consent were included in analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Versed | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 22 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.59 (0.9) | 3.45 (1.4) | 3.52 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Score From the Modified Yale Preoperative Anxiety Scale
Description: The modified Yale preoperative scale consists of 5 categories (activity, vocalizations, emotional expressivity, state of apparent arousal, and use of parents). Four of the five categories are scored between 1-4 points and one of the categories is scored from 1-6 points. The scores are divided by their number of possible points in their respective category and multiplied by 20 to get the final anxiety score which ranges from 20 to 100. Low numbers represent low anxiety and higher numbers represent high anxiety.
Time Frame: Waiting room, before catheterization, and after catheterization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Versed | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  Waiting Room | 30.80 (13.97) | 25.72 (3.47)
  Before catheterization | 44.51 (20.68) | 57.55 (29.34)
  After catheterization | 79.01 (19.26) | 81.39 (29.86)

2. Secondary Outcome: Anxiety Score From the State-Trait Anxiety Inventory
Description: The State-Trait anxiety inventory is consists of 20 questions on a 4-point force-choice Likert-type response scales (scores 0 - 3). The 20 questions are summed together for final score. The score can range from 0 to 60 with higher scores representing higher levels of anxiety. This questionnaire was used to evaluate the anxiety level of the parents of the children who randomized to versed or placebo.
Time Frame: At the time of the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Versed: Parents of patients who were given oral midazolam prior to undergoing the VCUG.
- Placebo: Parents of patients who were given oral placebo prior to undergoing the VCUG.
Arm/Group | Versed | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  Mothers | 10.07 (15.26) | 11.72 (13.75)
  Fathers | 13.54 (12.50) | 5.00 (7.35)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Versed | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes